CLINICAL TRIAL: NCT05808569
Title: Evaluating Breast Cancer Patients Modesty During Radiotherapy. A Multicentric Study
Acronym: MODESTY
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 3049
Record Dates: First submitted 2023-03-02; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer patients undergoing radiotherapy in adjuvant setting
  Interventions: Behavioral: Test

INTERVENTIONS:
Behavioral: Test — A specific self-test composed by 16 questions , will be administered to BC patients undergoing adjuvant RT.

SUMMARY:
Patients affected by breast cancer undergo radiotherapy with bare chest and can therefore live the moments in which they undress in front of the radiation therapy technologists (RTTs) in charge of their treatment as an extremely embarrassing one.

Furthermore, for some of these patients the relationship with their bodies has indeed changed since surgery (i.e. mutilations, scars), particularly for specific age or socio-economic groups. In this context, sub-standard care in maintaining modesty during breast cancer radiotherapy has been reported in literature, even if poorly studied. Aim of this multicentric observational study is to describe how modesty is perceived by patients undergoing radiotherapy for breast cancer.

ELIGIBILITY:
Inclusion criteria

* Patients undergoing adjuvant radiotherapy for breast cancer
* Able to understand and sign informed consent

Exclusion criteria

* Patients with inadequate linguistic abilities and inability to express informed consent
* Patients denying informed consent
* Patients receiving palliative treatments
* Patients affected by major psychiatric disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients undergoing adjuvant radiotherapy for breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 537 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Primary aim of this study is to identify patients perception of modesty during RT for breast cancer through the use of a dedicated 16 items questionnaire validated in a Delphi consensus for the purposes of this study | 1-5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario "A.Gemelli" IRCCS, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No